CLINICAL TRIAL: NCT01745289
Title: Long-term Anastrozole Versus Tamoxifen Treatment Effects (LATTE)
Brief Title: Long-term Anastrozole Versus Tamoxifen Treatment Effects
Acronym: LATTE
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00050408
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Survival; Recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Established in 2010, the Long-term Anastrozole vs Tamoxifen Treatment Effects (LATTE) observational study aims to collect vital long-term safety and efficacy data on anastrozole and tamoxifen, drugs that were taken by post-menopausal women as part of the Anastrozole Tamoxifen Alone or in Combination (ATAC) trial. ATAC was a crucial breast cancer trial evaluating the use of aromatase inhibitors (AIs) in the adjuvant setting, with a median follow-up of over 10 years. The ATAC trial assessed the safety and efficacy of anastrozole+placebo, tamoxifen+placebo and anastrozole+tamoxifen in postmenopausal women undergoing treatment for invasive primary breast cancer

DETAILED DESCRIPTION:
The LATTE study aims to collect further follow-up information on a maximum of 2200 UK eligible patients, who were randomised to the monotherapy arms (anastrozole or tamoxifen) in the ATAC trial. The LATTE study also aims to collect follow-up information on as many eligible patients as possible in international sites in the EU, US and Australia/New Zealand who were randomised to the monotherapy arms (anastrozole or tamoxifen) in the ATAC trial. The study's primary objective is to provide additional efficacy and safety data on time to recurrence of breast cancer and death after recurrence. The secondary objectives include time to distant recurrence, cancer-specific survival, new breast primaries, other cancers, ischaemic cardiac and cerebrovascular events and hip (and other) fractures. Participants will be followed-up annually until at least 15 years median follow-up.

In 2010, results from 10-year follow-up from ATAC demonstrated that there is long-term superiority of anastrozole over tamoxifen as initial adjuvant therapy for post-menopausal women with hormone-sensitive early breast cancer. This paper demonstrated that there were significantly lower rates of local and distant recurrence, as well as reduced contralateral breast cancer in patients treated with anastrozole. However, in 2016 a recent preliminary analysis of the LATTE study demonstrated that the benefits of anastrozole do not continue long-term after 10 years in terms of reduced recurrence rates. The results also suggested that there was a larger reduction of new contralateral tumours with tamoxifen. However, the preliminary analysis was limited in that there was limited data with possible under reporting of vital events inked to the safety and efficacy endpoints; this therefore may diminish the effect of anastrozole. Queen Mary University of London (QMUL) therefore require extended cohort events, obtainable from HES, cancer registration and mortality data in order to conclude the long-term safety of either intervention. QMUL will then be able to integrate the pseudonymised LATTE data with the ATAC data sets in order to perform an analysis of the overall 20-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* patients randomised to one of the monotherapy arms in the ATAC Trial
* alive at 10 years follow-up

Exclusion Criteria:

* patients who have withdrawn consent to participate in the ATAC Trial or this study
* where the LATTE Executive Committee determines that there is no possibility of obtaining follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with breast cancer who were randomised to receive either anastrozole or tamoxifen in the ATAC Trial and not known to have died or withdrawn consent before April 1st 2009 over the age of 18, living in the United States are eligible for LATTE.
Sampling Method: Non-Probability Sample
Enrollment: 2671 (Actual)
Dates: Start 2010-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | LATTE particpants who are 10 years post treatment will be followed for 5 years for the purpose of this study.
  Time to recurrence of breast cancer in the post 10 year period (defined as the earliest of local or distant recurrence, new primary breast cancer, or death)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smith, PhD, Principal Investigator — American Cancer Society, Inc.; Aman Buzdar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Queen Mary University of London, London, England, United Kingdom

REFERENCES:
- [Background] Cuzick J, Sestak I, Baum M, Buzdar A, Howell A, Dowsett M, Forbes JF; ATAC/LATTE investigators. Effect of anastrozole and tamoxifen as adjuvant treatment for early-stage breast cancer: 10-year analysis of the ATAC trial. Lancet Oncol. 2010 Dec;11(12):1135-41. doi: 10.1016/S1470-2045(10)70257-6. Epub 2010 Nov 17. PMID 21087898
- [Background] Allawi Z, Cuzick J, Baum M; ATAC/LATTE investigators. Does trauma or an intercurrent surgical intervention lead to a short-term increase in breast cancer recurrence rates? Ann Oncol. 2012 Apr;23(4):866-9. doi: 10.1093/annonc/mdr316. Epub 2011 Jul 15. PMID 21765042